CLINICAL TRIAL: NCT02552654
Title: Cortisol and the Formation of Intrusive Memories: An Experimental Approach With a Trauma Film Paradigm
Brief Title: Cortisol and the Formation of Intrusive Memories
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Felicitas Rombold, Dipl.-Psych., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Rombold_02
Record Dates: First submitted 2015-09-16; First posted 2015-09-17 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Intrusive Memories
MeSH Terms: interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrocortisone and Stress Film (Experimental): Administration of 10mg hydrocortisone before the trauma film.
  Interventions: Behavioral: Stress Film; Drug: Hydrocortisone
- Placebo and Stress Film (Experimental): Administration of placebo before the trauma film.
  Interventions: Behavioral: Stress Film; Drug: Placebo

INTERVENTIONS:
Behavioral: Stress Film — Film scene with severe physical and sexual violence.
Drug: Hydrocortisone — 10mg
  Arms: Hydrocortisone and Stress Film
Drug: Placebo
  Arms: Placebo and Stress Film

SUMMARY:
Intrusive memories of traumatic events are core features of posttraumatic stress disorder (PTSD) but little is known about the neurobiological formation of intrusions. The aim of this study was to determine whether cortisol levels during an intrusion-inducing stressor influence subsequent intrusive memories.

DETAILED DESCRIPTION:
The investigators conducted an experimental, double-blind, placebo-controlled study in 60 healthy women. Prior to watching an established trauma film paradigm that induces short lasting intrusions, participants received a single dose of either 10 mg hydrocortisone or placebo. The number of consecutive intrusions of the trauma film, the mean vividness of the intrusions and the mean degree of distress evoked by the intrusions were assessed during the following seven days. Salivary cortisol and alpha-amylase were collected at seven time points prior to, and after the trauma film.

ELIGIBILITY:
Inclusion Criteria:

* healthy participants
* German on a native level

Exclusion Criteria:

* former or present DSM IV Axis I disorders
* physical illnesses
* any medication intake (except oral contraceptive)
* history of sexual abuse or rape
* pregnancy or lactation period

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of intrusive memories | seven consecutive days
  Measured with an intrusion diary

SECONDARY OUTCOMES:
Vividness of intrusive memories | seven consecutive days
  Measured with an intrusion diary
Degree of distress of intrusive memories | seven consecutive days
  Measured with an intrusion diary

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Roepke, Study Director — Charite University, Berlin, Germany